CLINICAL TRIAL: NCT06239376
Title: The Effectiveness of the Two Different Endometrial Preparation Regimes for Frozen Embryo Transfer in Patients With Adenomyosis
Brief Title: Artificial Cycle With or Without GnRH Agonist Pre-treatment for Frozen Embryo Transfer in Adenomyosis Patients
Acronym: FET-ADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/23/DD-BVMD
Record Dates: First submitted 2023-12-18; First posted 2024-02-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Adenomyosis; IVF; Frozen Embryo Transfer
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH agonist + Letrzole - Artificial Cycle (Active Comparator): Pre-treatment includes two doses of 3.75 mg GnRH agonist (Diphereline®, Ipsen, France) on days 2-4 of the menstrual cycle and 28 days later, along with daily 2.5 mg Letrozole (Femara®, Novartis, Switzerland) starting from the first agonist injection.
  Endometrial preparation in an artificial cycle begins 28 days after the second agonist injection. Patients will take 6 mg/day of oral estradiol valerate (Valiera; Abbott) at least 9 days before initiating progesterone. Endometrial thickness is monitored starting on the 10th day. When it reaches ≥7 mm, 400 mg twice times a day of vaginal progesterone (Cyclogest®, Actavis, UK) is initiated. Embryo transfer aligns with progesterone initiation, taking the embryo's stage into account. Luteal phase support comprises oral estradiol valerate 4 mg/day and vaginal progesterone 400 mg twice times a day until the 7th week of gestational age (GA), followed by progesterone alone at 400 mg twice times a day up to the 12th week of GA.
  Interventions: Procedure: GnRHa+AI - AC
- Artificial Cycle (Active Comparator): The endometrium will be prepared using oral estradiol valerate (Valiera; Abbott) 6 mg/day starting from the 2nd to the 4th day of the menstrual cycle. The endometrial thickness will be monitored from day 10th onwards, and vaginal progesterone (Cyclogest®; Actavis) 400 mg twice times a day will be initiated when endometrial thickness reaches ≥7 mm. Estradiol exposure must last for at least 9 days before progesterone administration. Embryo transfer will be scheduled by the time of the initiation of progesterone and embryo stages. Luteal phase support comprises oral estradiol valerate 4 mg/day and vaginal progesterone 400 mg twice times a day until the 7th week of gestational age (GA), followed by progesterone alone at 400 mg twice times a day up to the 12th week of GA.
  Interventions: Procedure: Artificial cycle

INTERVENTIONS:
Procedure: GnRHa+AI - AC — Pre-treatment includes two doses of 3.75 mg GnRH agonist (Diphereline®, Ipsen, France) on days 2-4 of the menstrual cycle and 28 days later, along with daily 2.5 mg Letrozole (Femara®, Novartis, Switzerland) starting from the first agonist injection.
  Endometrial preparation in an artificial cycle begins 28 days after the second agonist injection. Patients take 6 mg/day of oral estradiol valerate (Valiera; Abbott) at least 9 days before progesterone. Endometrial thickness is monitored starting on the 10th day. When it reaches ≥7 mm, 400 mg twice times a day of vaginal progesterone (Cyclogest®, Actavis, UK) is initiated. Embryo transfer aligns with progesterone initiation, taking the embryo's stage into account. Luteal phase support comprises oral estradiol valerate 4 mg/day and vaginal progesterone 400 mg twice times a day until the 7th week of gestational age (GA), followed by progesterone alone at 400 mg twice times a day up to the 12th week of GA.
  Other Names: DR-AC
  Arms: GnRH agonist + Letrzole - Artificial Cycle
Procedure: Artificial cycle — The endometrium will be prepared using oral estradiol valerate (Valiera; Abbott) 6 mg/day starting from the 2nd to the 4th day of the menstrual cycle. The endometrial thickness will be monitored from day 10th onwards, and vaginal progesterone (Cyclogest®; Actavis) 400 mg twice times a day will be initiated when endometrial thickness reaches ≥7 mm. Estradiol exposure must last for at least 9 days before progesterone administration. Embryo transfer will be scheduled by the time of the initiation of progesterone and embryo stages. Luteal phase support comprises estradiol 4 mg/day and vaginal progesterone 400 mg twice times a day until the 7th week of gestational age (GA), followed by progesterone alone at 400 mg twice times a day up to the 12th week of GA.
  Other Names: AC
  Arms: Artificial Cycle

SUMMARY:
This randomized clinical trial aims to assess the comparative effectiveness of two distinct endometrial preparation protocols for frozen embryo transfer (FET) among women with adenomyosis undergoing IVF/ICSI. Specifically, it seeks to address the following key questions:

1. Does the protocol involving the combination of GnRH agonist and letrozole for down regulation with exogenous steroids (GnRHa+AI - AC) result in a higher live birth rate compared to the use of exogenous steroids alone (AC) in women with adenomyosis undergoing frozen embryo transfer?
2. What are the common side effects of the GnRHa+AI - AC regimen?

Eligible participants will undergo screening before endometrial preparation for FET, following which they will be randomly assigned to one of two groups: GnRHa+AI - AC or AC. In the GnRHa+AI - AC group, participants will be pre-treated with GnRH agonist and letrozole two months before endometrial preparation. After this period, participants will return for endometrial preparation, and any side effects resulting from the down regulation will be evaluated. In contrast, the AC group will receive standard treatment.

DETAILED DESCRIPTION:
* Adenomyosis is a benign gynecological disease in which the endometrial stroma invades the uterine myometrium. Adenomyosis affects approximately 10% of women of reproductive age. There are several hypothetical mechanisms in adenomyosis-associated infertility, including dysregulations of the myometrial architecture and function, chronic inflammation, presence of local oxygen, and altered endometrial function, which can cause implantation failure. The abnormal presence of endometrial tissue composed of glands and stroma impacts uterine smooth muscle's regular contractile function and peristalsis, resulting in menometrorrhagia, infertility, and adverse obstetric consequences. There is currently no consensus on the optimal protocol for endometrial preparation in this population, and a lack of data on this issue. Current protocols include routine protocols with or without the pre-treatment of GnRH agonist. However, it is still controversial whether GnRH agonist down-regulation can help patients with adenomyosis have better reproductive outcomes. To our knowledge, there have not been any randomized controlled trials to investigate the effectiveness of the protocols used for endometrial preparation in women with adenomyosis undergoing frozen embryo transfer.
* This will be a superiority-designed randomized clinical trial.
* This trial will be conducted at My Duc Hospital, Ho Chi Minh City, Vietnam. Potentially eligible women will be provided information about the trial as long as their stimulation cycles are initiated.
* Screening for eligibility will be performed by treating physicians on days 2nd - 4th of the menstrual cycle in the subsequent frozen embryo transfer cycles. Patients will be provided a copy of the informed consent documents. Written informed consent will be obtained from all women by the investigator before enrollment.
* Women will be randomized (1:1) to either AC (artificial cycle) or GnRHa+AI - AC (Down-Regulation with GnRH agonist and Letrozole combined with artificial cycle) protocols using block randomization with a variable block size of 4, 6, using HOPE Epi with a computer-generated random list.
* Artificial cycle (AC): the endometrium will be prepared using oral estradiol valerate (Valiera; Abbott) 6 mg/day starting from the second or fourth day of the menstrual cycle (5). The endometrial thickness will be monitored from the tenth day of estradiol-priming onwards, and vaginal progesterone (Cyclogest®; Actavis) 400 mg twice times a day will be initiated when endometrial thickness reaches 7 mm or more and received oestradiol valerate for at least nine days.

Embryo transfer will be scheduled by the time of the initiation of progesterone and embryo stages. Hormonal support will consist of oral estradiol valerate 4 mg/day and vaginal progesterone (Cyclogest®; Actavis) 400 mg twice times a day until the 7th week of gestation. Subsequently, progesterone alone (Cyclogest®; Actavis) at 400 mg twice times a day will be continued for luteal phase support until the 12th week of gestation.

- GnRH agonist + Letrozole - Artificial cycle protocol (GnRHa+AI - AC):

* Pre-treatment with GnRH agonist: GnRHa (Triptorelin - Diphereline®, Ipsen, France) will be injected at a dose of 3.75 mg on days 2nd - 4th of menstruation. In addition to GnRHa administration duration, the patients will be indicated letrozole 2.5 mg daily (Femara®, Novartis, Switzerland) to prevent the estradiol flare-up effect from the day of GnRH agonist injection. Repeat the same regimen for the second time 28 days after the first injection of GnRH agonist.
* After 55 days of Down Regulation with GnRH agonist, before starting the artificial cycle protocol for endometrial preparation, estradiol serum level will be tested before endometrial preparation.
* Endometrial preparation with AC protocol will be started 28 days after the second injection of GnRH agonist, as described previously

Frozen embryo transfer:

A maximum of 2 cleavage-stage embryos or 1 blastocyst will be thawed on the day of embryo transfer, three or five days after the start of progesterone. Two hours after thawing, surviving embryos will be transferred into the uterus under ultrasound guidance using a soft uterine catheter (Gynétics®, Belgium).

- Future babies' health evaluation and cost-effectiveness analysis will also be performed separately.

ELIGIBILITY:
Inclusion Criteria:

* Confirm diagnosis with adenomyosis by using transvaginal ultrasonography (MUSA consensus) and/or pelvic magnetic resonance imaging.
* Age between 18 - 42
* Undergo less or equal to three previous IVF cycles
* Indicate for frozen embryo transfer
* Agree to have not more than two day-3 embryo or one blastocyst (day-5 and day-6) transferred
* Not participating in any other study

Exclusion Criteria:

* Embryos from IVM cycle
* Having uterine or adnexal abnormalities (e.g., intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus; unremoved hydrosalpinx, endometrial polyp, submucosal leiomyoma, or leiomyoma with endometrial cavity distortion)
* Having contraindications for exogenous hormones administration: breast cancer, risks of venous thromboembolism
* Embryos from the oocyte donation cycle.
* Patients with a history of GnRH injection within three months, measured from the last GnRHa injection to the study screening date.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after one frozen embryo transfer cycle | At 22 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown

SECONDARY OUTCOMES:
Cancellation rate | At 3 weeks from the start of artificial cycle
  Cancellation due to: thin endometrium (thickness <7mm after ≥21 days using oral estradiol valerate), endometrial cavity fluid, functional cyst (homogeneous anechoic cyst with d ≥14 mm present after 10 days using estradiol valerate), or has side effects(Cluster headache, mood swing, abnormal uterine bleeding, nausea, vomit, VTE, stroke)
Hypoestrogenic side effects | At 8 weeks from the start of the first dose of 3.75 mg GnRH agonist
  Side effects include hot flushes, bone loss, vaginal dryness, decreased libido, unpredictable mood changes, and headache.
Classification of adenomyosis | during ultrasound procedure
  The classification of adenomyosis under ultrasound scan according to MUSA criteria
Differentiation of adenomyosis | during ultrasound procedure
  The differentiation of adenomyosis under ultrasound scan according to MUSA criteria
Positive pregnancy test | At 2 weeks after embryo placement
  Serum ß-hCG ≥25mIU/mL
Implantation rate | At 3 weeks after embryo placement
  Implantation rate is explained as the number of gestational sacs per number of embryos transferred.
Clinical pregnancy | At 5 weeks after embryo placement
  diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more after the onset of the last menstrual period. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy.
Ectopic pregnancy | At 7 weeks of gestation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualisation, or histopathology
Ongoing pregnancy | At 10 weeks after embryo placement
  Having at least one gestational sac on ultrasound at 12 weeks' gestation with heart beat activity
Miscarriage | before 22 completed weeks of gestational age
  The spontaneous loss of an intra-uterine pregnancy before 22 completed weeks of gestational age
Venous thromboembolism relating to medication | From the start of treatment up to 10 weeks of gestation
  Venous thromboembolism is diagnosed after clinical examination, ultrasound scan and blood test
Preterm delivery | At 22, 28, 32 weeks and 37 weeks of gestation
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Gestational diabetes mellitus | At 24 to 28 weeks of gestation
  GDM is diagnosed using a 75g oral glucose tolerance test
Hypertension in pregnancy | after 20 weeks of gestation or beyond
  Pregnancy-induced hypertension, pre-eclampsia, eclampsia and HELLP syndrome
Major congenital abnormalities | At birth
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally, at birth or later in life. Congenital anomalies can be caused by single gene defects, chromosomal disorders, multifactorial inheritance, environmental teratogens and micronutrient deficiencies. The time of identification should be reported. Any congenital anomaly will be included as followed definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
Birth weight | At the time of delivery
  Weight of singletons and twins
Low birth weight | At the time of delivery
  Weight < 2500 gm at birth
Very low birth weight | At the time of delivery
  Weight < 1500 gm at birth
High birth weight | At the time of delivery
  Weight 4000 gm or 4500 gm at birth
Very high birth weight | At the time of delivery
  Weight over than 4.500 g for women with diabetes, and a threshold of 5000 g for women without diabetes
Admission to NICU | At birth
  The admittance of the newborn to NICU
Multiple pregnancy | At 6 to 8 weeks' gestation
  ≥2 gestational sac at early pregnancy ultrasound
Multiple delivery | At 22 weeks' gestation
  Birth of more than one baby beyond 22 weeks
Still birth | At 20 weeks' gestation
  The death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles.
Neonatal mortality | within 28 days of birth
  Death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between eight and 28 days after delivery
Direct costs to live birth | At the time of delivery
  Total direct cost to have a live birth after embryo transfer. Direct cost include medical consultations, ovulation stimulation drugs, laboratory and embryology services, ultrasound scanning, medical procedures such as oocyte retrieval and embryo transfer, hospital charges, nursing and counselling services and administrative and overhead charges (Mark P. Connolly et al., 2010). Cost data will be collected for a supplementary analysis and will be reported in a separated paper.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zondervan KT, Becker CM, Missmer SA. Endometriosis. N Engl J Med. 2020 Mar 26;382(13):1244-1256. doi: 10.1056/NEJMra1810764. No abstract available. PMID 32212520
- [Background] Szubert M, Kozirog E, Olszak O, Krygier-Kurz K, Kazmierczak J, Wilczynski J. Adenomyosis and Infertility-Review of Medical and Surgical Approaches. Int J Environ Res Public Health. 2021 Jan 30;18(3):1235. doi: 10.3390/ijerph18031235. PMID 33573117
- [Background] Antero MF, Ayhan A, Segars J, Shih IM. Pathology and Pathogenesis of Adenomyosis. Semin Reprod Med. 2020 May;38(2-03):108-118. doi: 10.1055/s-0040-1718922. Epub 2020 Oct 20. PMID 33080632
- [Background] Mumusoglu S, Polat M, Ozbek IY, Bozdag G, Papanikolaou EG, Esteves SC, Humaidan P, Yarali H. Preparation of the Endometrium for Frozen Embryo Transfer: A Systematic Review. Front Endocrinol (Lausanne). 2021 Jul 9;12:688237. doi: 10.3389/fendo.2021.688237. eCollection 2021. PMID 34305815
- [Background] Zhang Y, Fu X, Gao S, Gao S, Gao S, Ma J, Chen ZJ. Preparation of the endometrium for frozen embryo transfer: an update on clinical practices. Reprod Biol Endocrinol. 2023 Jun 8;21(1):52. doi: 10.1186/s12958-023-01106-5. PMID 37291605
- [Background] Harmsen MJ, Van den Bosch T, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Hehenkamp WJK, Groenman F, De Bruyn C, Rasmussen C, Lazzeri L, Jokubkiene L, Jurkovic D, Naftalin J, Tellum T, Bourne T, Timmerman D, Huirne JAF. Consensus on revised definitions of Morphological Uterus Sonographic Assessment (MUSA) features of adenomyosis: results of modified Delphi procedure. Ultrasound Obstet Gynecol. 2022 Jul;60(1):118-131. doi: 10.1002/uog.24786. PMID 34587658